CLINICAL TRIAL: NCT05434052
Title: Turkish Adaptation, Validity and Reliability of Community Integration Questionnaire-Revised (CIQ-R)
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research Assistant, Istanbul Medeniyet University
Other Study IDs: CIQ-R
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Community Integration
Keywords: stroke; social networking; social participation; community integration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patients: The aim of this study is to adapt the Community Integration Questionnaire-Revised (CIQ-R)scale to Turkish society in stroke patients and to make its validity and reliability in Turkish.
  Interventions: Other: Turkish Validity and Reliability of The CIQ-R Scale

INTERVENTIONS:
Other: Turkish Validity and Reliability of The CIQ-R Scale — The aim of this study is to adapt the Community Integration Questionnaire-Revised (CIQ-R)scale to Turkish society and to make its validity and reliability in Turkish. It has 18 questions. This study will be conducted with stroke patients. The patients will be sought to answer questionnaires during regular rehabilitation sessions.

SUMMARY:
The aim of this study is to adapt the Community Integration Questionnaire-Revised (CIQ-R) scale to Turkish society and to make its validity and reliability in Turkish. The CIQ-R scale developed by Callaway et al assesses home integration, social integration, productivity, and electronic social networking in neurological diseases. It has 18 questions. This study will be conducted with stroke patients. The patients will be sought to answer questionnaires during regular rehabilitation sessions. 130 participants will be included in the study. In order to evaluate the validity of the CIQ-R, the Mini Mental State Examination (MMSE), which can evaluates general cognitive functioning and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion.

The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. If the developer of the scale, Callaway and Willer approves the translation of the scale, participants will be recruited for the study. In the pre-trial phase, a reassessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of CIQ-R will be able to be modified. The data of CIQ-R are collecting through face-to-face when the patients came to the rehabilitation center. 145 participants will be included in the study.

In order to evaluate the validity of the CIQ-R, the Mini Mental State Examination (MMSE), which can evaluates general cognitive functioning and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

Patients with

* duration of hemiplegia ≤ 3 year
* able to speak and read Turkish
* those with a Mini Mental State Examination score of 24 and above

Exclusion Criteria: Patients with

* communication or cognitive problems,
* aphasia and speech disorders
* unstable medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients who are aged 18-65 years with duration of hemiplegia ≤ 3 years and able to speak and read Turkish.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
community integration | baseline
  community integration will be assessed with the Community Integration Questionnaire-Revised (CIQ-R) scale. It consists of 18 items in total. Each item is scored on a scale of 0-2 includes four sub-categories: Home Integration (HI), Social Integration (SI), Productivity (P), and Electronic Social Network (ESN).
  The total score is the calculated sum of 18 items. The minimum score is 0 and the maximum score is 35 points. Higher scores indicate a high level of community integration which means better community integration.
Cognitive function | baseline
  The Mini-Mental State Examination (MMSE), which is a widely used cognitive assessment questionnaire is quite short. It evaluates general cognitive functioning (especially in the left cerebral hemisphere) and ranged from 0 to 30 points. According to the scale results; It is accepted that there is severe cognitive influence between 0-17 points, moderate cognitive influence between 18-23 points, and no cognitive influence between 24-30 points. Higher scores mean better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)